CLINICAL TRIAL: NCT04046263
Title: Effect of Velphoro on Serum Phosphate and Albumin in Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1027
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Results first posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Peritoneal Dialysis Complication; Hyperphosphatemia; Hypoalbuminemia
MeSH Terms: conditions — Hyperphosphatemia; Hypoalbuminemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention (Experimental): Open-label, one arm study. Patients receive sucroferric oxyhydroxide three times daily and dose is titrated to keep serum phosphate at goal.
  Interventions: Drug: Sucroferric Oxyhydroxide Chewable Tablet

INTERVENTIONS:
Drug: Sucroferric Oxyhydroxide Chewable Tablet — Patients will be started on 1 tablet three times daily with meals and the dose will be titrated monthly in increments of 500mg (1 tablet) per day until serum phosphate is at goal

SUMMARY:
Prospective pilot study to determine if changing the phosphate binder to sucroferric oxyhydroxide for for 6 months improves disordered mineral metabolism and nutrition status in peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* On peritoneal dialysis at least 3 months with a Kt/V of ≥ 1.7
* Use of Automated Peritoneal Dialysis
* Serum phosphate > 5.5 mg/dL or <5.5 mg/dL on a binder other than velphoro
* Serum albumin ≤ 3.7 g/dL
* Able to provide consent
* Ability to complete self-reported questionnaire

Exclusion Criteria:

* Inadequate dialysis
* Current use of sucroferric oxyhydroxide
* Significant comorbid conditions that lead the investigator to conclude that life expectancy is less than 6 months
* Active malignancy
* Recent episode of peritonitis
* Pregnancy or planning to become pregnant
* Anticipated kidney transplantation within 6 months
* Factors judged to limit adherence to interventions
* Known adverse side effect to sucroferric oxydroxide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kendrick, MD, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study deidentified data will be available to other researchers
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available at the completion of the study. Researchers must obtain PI approval

REFERENCES:
- [Derived] Perez L, You Z, Teitelbaum I, Andrews ES, Reddin R, Ramirez-Renteria L, Wilson G, Kendrick J. A 6-Month clinical practice pilot study of sucroferric oxyhydroxide on nutritional status in patients on peritoneal dialysis. BMC Nephrol. 2022 Jul 9;23(1):245. doi: 10.1186/s12882-022-02878-5. PMID 35810296

RESULTS

PARTICIPANT FLOW:
Groups:
- Sucroferric Oxyhydroxide: Open-label, one arm study. Patients receive sucroferric oxyhydroxide three times daily and dose is titrated to keep serum phosphate at goal.
  Sucroferric Oxyhydroxide Chewable Tablet: Patients will be started on 1 tablet three times daily with meals and the dose will be titrated monthly in increments of 500mg (1 tablet) per day until serum phosphate is at goal
Period: Overall Study
Arm/Group | Sucroferric Oxyhydroxide
Started | 17
Completed | 12
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Serum Phosphate at Baseline
Description: Serum phosphate at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention
Number analyzed (Participants) | 17
mg/dL | 7.47 (1.76)

2. Primary Outcome: Serum Phosphate at 6 Months
Description: Serum phosphate at end of study (6 months)
Time Frame: 6 months
Population: Outcome measure data could not be collected for all participants at the 6 month timepoint due to some participants discontinuing the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention
Number analyzed (Participants) | 12
mg/dL | 5.69 (1.17)

3. Secondary Outcome: Serum Albumin
Description: Changes in serum albumin from baseline to 6 months
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Intervention
Number analyzed (Participants) | 17
g/dL
  Baseline | 3.49 (0.37)
  6 Months: number analyzed (Participants) | 12
  6 Months | 3.50 (0.27)

4. Secondary Outcome: Serum FGF23
Description: Change in serum FGF23 from baseline to 6 months
Time Frame: 6 months
Population: This outcome measure could not be collected due to unforeseen changes in the study capability caused by the COVID-19 public health crisis.
Arm/Group | Intervention
Number analyzed (Participants) | 0

5. Secondary Outcome: Serum PTH
Description: Change in serum PTH (perathyroid hormone) from baseline to 6 months
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: picograms/mL
Arm/Group | Intervention
Number analyzed (Participants) | 17
picograms/mL
  Baseline | 416 [292 to 631]
  6 Months: number analyzed (Participants) | 12
  6 Months | 361 [237 to 540]

6. Secondary Outcome: Serum Prealbumin
Description: Change in prealbumin from baseline to 6 months
Time Frame: 6 months
Population: as for outcome 4
Arm/Group | Intervention
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 2/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 9/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=17)
Death (Cardiac disorders) | 2 (2) — 2 participants died, likely due to COVID-19. Was determined not to be study related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=17)
GI symptoms (Gastrointestinal disorders) | 9 (9) — includes common GI symptoms such as nausea & vomiting.

LIMITATIONS AND CAVEATS:
Study sample size is very small and there is no control group. This was due to complications that arose from the COVID-19 public health crisis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT04046263/Prot_SAP_000.pdf